CLINICAL TRIAL: NCT02473627
Title: A PHASE 1, OPEN-LABEL, CROSS-OVER, FIXED SEQUENCE STUDY TO EVALUATE THE EFFECT OF MULTIPLE DOSES OF DS-1971A ON THE SINGLE DOSE PHARMACOKINETICS OF PROBE SUBSTRATES FOR CYP2B6, CYP2C8, CYP2C9, CYP2C19 AND CYP3A4 ENZYMES IN HEALTHY MALE AND FEMALE SUBJECTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DS1971-A-E105
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Pharmacokinetics
MeSH Terms: interventions — DS-1971a; Midazolam; Omeprazole; Pioglitazone; Tolbutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1 (Experimental): Period 1 Day 1: single oral dose of 2.5 mg midazolam hydrochloride Day 2: single oral cocktail dose of 20 mg omeprazole, 15 mg pioglitazone hydrochloride, 500 mg tolbutamide and 150 mg bupropion
  Interventions: Drug: midazolam hydrochloride; Drug: Omeprazole; Drug: Pioglitazone hydrochloride; Drug: Buproprion; Drug: Tolbutamide
- Period 2 (Experimental): Period 2 Days 1 through 12 repeated doses of 400 mg DS-1971a administered orally bid .
  On the days listed below, each probe substrate(s) will be coadministered with the morning dose of DS 1971a:
  Day 8: single oral dose of 2.5 mg midazolam hydrochloride Day 9: single oral cocktail dose of 20 mg omeprazole, 15 mg pioglitazone hydrochloride, 500 mg tolbutamide and 150 mg bupropion
  Interventions: Drug: DS-1971a; Drug: midazolam hydrochloride; Drug: Omeprazole; Drug: Pioglitazone hydrochloride; Drug: Buproprion; Drug: Tolbutamide

INTERVENTIONS:
Drug: DS-1971a — 200mg tablet
  Arms: Period 2
Drug: midazolam hydrochloride — 2.5mg oromucosal liquid
Drug: Omeprazole — 20mg gastro-resistant capsule
Drug: Pioglitazone hydrochloride — 15mg tablet
Drug: Buproprion — 150mg Prolonged release tablet
Drug: Tolbutamide — 500mg tablet

SUMMARY:
This is an open-label, cross-over, fixed-sequence study. All subjects will receive the same treatment in two study periods. The study is designed to test whether DS-1971a has any effect on the activity of various enzymes involved in the metabolism of medicines, using test medications. These will be given without and then with DS-1971a to see if DS-1971a has any effect on the blood levels of the test medicines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 65 years, inclusive.
* Be in good general health as determined by medical history, physical examination and Screening investigations, and be taking no regular medication.
* A body mass index (BMI) in the range 18 to 30 kg/m2, inclusive, and weighing between 50 and 100 kg, inclusive. BMI is calculated as weight [kg]/(height [m])*2.
* Female subjects must be of nonchildbearing potential as follows:

Must be postmenopausal (the last menstrual period was at least 12 months before Screening, and a follicle stimulating hormone [FSH] test at Screening confirms postmenopausal status); or Must be surgically sterile having undergone hysterectomy, bilateral oophorectomy, bilateral salpingectomy and/or bilateral tubal ligation.

* Willing to comply with all study restrictions, including the use of contraception, concomitant medication and dietary and lifestyle restrictions.
* Possessing sufficient intelligence to understand the nature of the study and any hazards of participating in it, and the ability to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire study.
* Have given written consent to participate after reading the ICF, and after having the opportunity to discuss the study with the Investigator or his/her delegate.
* Have given written consent to have his/her data entered into The Overvolunteering Prevention System.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG findings or laboratory values that could interfere with the objectives of the study or the safety of the subject.
* Presence of history of acute or chronic illness, including (but not limited to) liver or kidney disease, hypertension, seizures, or any known impairment of endocrine, or other specific body-organ dysfunction.
* Presence or history of severe adverse reaction to any medicine.
* Presence or history of malignant disease.
* Acute or chronic infectious disease, including human immunodeficiency virus (HIV), hepatitis B virus or C virus (HCV) infection.
* Surgery (eg, stomach bypass) or medical condition that might affect absorption of medicines.
* Significant illness within 4 weeks before the dose of study medication.
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months, or unwilling to abstain from participating in other clinical trials during the study and for 3 months after receipt of study medication.
* Participation in another clinical study with DS-1971a.
* Blood pressure (BP) and heart rate in semisupine position at the Screening examination outside the ranges 90 to 140 mmHg systolic, 40 to 90 mmHg diastolic; heart rate 40 to 100 beats/min. Subjects with Stage 1 hypertension (systolic 140 to 160 mmHg; diastolic 90 to 100 mmHg) may be enrolled provided they do not have evidence of end-organ damage, diabetes or a 10 year cardiovascular risk > 20%.
* Abnormal ECG waveform morphology at Screening that would preclude accurate measurement of the uncorrected QT interval (QT) duration.
* QT interval for heart rate corrected using Fridericia's formula (QTcF) interval duration > 430 msec for men or > 450 msec for women, obtained as an average from the measurements on duplicate Screening ECGs.
* Estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73 m*2 or an absolute creatinine value above the upper limit of the normal range. eGFR will be estimated at Screening using the Modification of Diet in Renal Disease (MDRD) equation.
* Poor metaboliser genotype status for CYP2C9 and CYP2C19 (Note: this exclusion criterion is to ensure that the study population is sensitive to a metabolic interaction).
* Use of any prescription medicine, over the counter (OTC) medications, herbal remedies (such as St John's Wort), or food known to be strong inhibitors or strong inducers of CYP enzymes (also known as CYP450 enzymes) during the 30 days before the dose of study medication; use of any other prescription or OTC medicine, including dietary supplements or herbal remedies, during the 7 days before the first dose of study medication.
* Consumption of certain foods or beverages before the dose and throughout the study period.
* Loss of more than 400 mL blood plasma, platelets or any other blood components during the 3 months before the first dose of study medication, or unwilling to abstain from doing so during the study and for 3 months after receipt of study medication.
* Abuse of drugs or alcohol in the past, or intake of more than 21 units of alcohol weekly (for men) or 14 units of alcohol weekly (for women).
* Use of tobacco products or nicotine containing products during the 3 months before the dose of study medication.
* Likely possibility that the subject will not cooperate with the requirements of the protocol.
* Objection by General Practitioner to subjects entering the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile for bupropion | Days 2-6 of Period 1 and Day 9-13 of Period 2
  Pharmacokinetic parameters (Cmax, tmax , AUC) for bupropion when administered without or with DS-1971a
Pharmacokinetic profile for pioglitazone | Days 2-4 of Period 1 and Days 9-11 of Period 2
  Pharmacokinetic parameters (Cmax, tmax , AUC) for pioglitazone when administered without or with DS-1971a
Pharmacokinetic profile for tolbutamide | Days 2-4 of Period 1 and Days 9-11 of Period 2
  Pharmacokinetic parameters (Cmax, tmax , AUC) for tolbutamide when administered without or with DS-1971a
Pharmacokinetic profile for omeprazole | Day 2 of Period 1 and Day 9 of Period 2
  Pharmacokinetic parameters (Cmax, tmax , AUC) for omeprazole when administered without or with DS-1971a
Pharmacokinetic profile for midazolam | Day 1 of Period 1 and Day 8 of Period 2
  Pharmacokinetic parameters (Cmax, tmax , AUC) for midazolam when administered without or with DS-1971a

SECONDARY OUTCOMES:
Pharmacokinetic profile of DS-1971a | Day 1, 3, 6, 8, 9, and 12
  PK parameters (Cmax , Ctrough , Cavg , tmax , AUC) of DS 1971a and its metabolites
Pharmacokinetic profile of metabolites of substrates | Days 1-6 of Period 1 and Days 8-13 of Period 2
  PK parameters (Cmax , tmax , AUC, metabolite/parent ratio) of metabolites of bupropion, omeprazole, tolbutamide, and midazolam
number and severity of Adverse Events | Day 0 - Week 9
  The number, severity, and percentage of subjects reporting Treatment Emergent Adverse Events (TEAEs) will be tabulated.

CONTACTS AND LOCATIONS:
Locations (1):
- London, United Kingdom